CLINICAL TRIAL: NCT05556707
Title: Symptom Clusters and Risk Factors of Patients Recovering From COVID-19 Caused by Omicron BA.2
Brief Title: Symptom Clusters and Risk Factors of COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2022-003-B
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; Patient Discharge; Symptoms and Signs
Keywords: COVID-19; patient discharge; symptoms and signs; sensation; nervous system; emotions; respiratory system; pain; nursing assessment; disease management
MeSH Terms: conditions — COVID-19; Signs and Symptoms; Neurologic Manifestations; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim and objectives: To clarify the types, composition, distribution characteristics and risk factors of symptom clusters experienced by discharged patients with COVID-19, to lay the foundation for effective symptom management.

Background: Even when patients recover from COVID-19 patients, the virus can still cause many long-term effects or complications.Therefore, it is crucial to assess the symptoms and influencing factors of discharged patients with COVID-19.

Design: Cross-sectional survey. Methods:The investigators used the Post Discharge Experience Assessment Questionnaire for COVID-19 Patients and the Post Discharge Symptom Experience Risk Factor Questionnaire for COVID-19 Patients were used.Stratified random sampling was used to conduct a cross-sectional survey of 384 patients in recovery from COVID-19.Exploratory factor analysis was used to determine the cluster of symptoms, and a binary logistic regression analysis was used to identify the risk factors associated with this symptom cluster.

DETAILED DESCRIPTION:
1. A Symptom Experience Assessment Questionnaire for COVID-19 patients after recovery; a self-designed symptom assessment tool. The questionnaire takes the Symptom Experience Model (Armstrong et al., 2003) as the theoretical framework, and combines it with a systematic review of COVID-19 symptoms of patients in recovery to form the entry pool. The questionnaire included twenty-four symptoms, and each symptom included three dimensions: frequency, severity, and distress. Each dimension was scored using Likert scales. Taking frequency as an example, zero represents "never happened" and 4 represents "always existed". Cronbach's α coefficient: 0.953, split half reliability: 0.949; KMO: 0.842; (Bartlett's Test of Sphericity) Sig is 0.
2. A questionnaire on risk factors of symptom experience of COVID-19 patients after recovery: a self-designed survey tool.The questionnaire is based on the Symptom Experience Model. In this model, sociodemographic characteristics, disease-related characteristics, and personal characteristics are taken to be the leading factors of symptom experience, and three factors jointly mediate the occurrence and development of symptom experience. Based on this, combined with the results of the literature analysis and the clinical experience in our team, the investigators developed a questionnaire on the factors that influence the experience of symptoms in COVID-19 patients after recovery This included three parts, (a) sociodemographic characteristics (age, marital status, educational background) (b) disease-related characteristics (length of hospitalization, days following discharge, retesting positive for COVID-19, chronic disease) (c) individual factors (the main ways of acquiring knowledge of COVID-19, authenticity of optimism, the degree to which work is affected by symptoms, satisfaction with daily life). Each item was scored by the Likert 5-level scoring method, with zero representing "never" and 4 representing "always".

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with COVID-19 who have been discharged from the hospital and clearly aware and able to communicate normally.

Exclusion Criteria:

* Patients who have not recovered or are still in the makeshift hospitals and those who refused to participate in the follow-up survey.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From March to May 2022, patients treated at Shanghai Xinguo Bo Makeshift Hospital and Renji Hospital, School of Medicine, Shanghai Jiaotong University, were selected as research participants.
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Post Discharge Experience Assessment Questionnaire for COVID-19 Patients and the Post Discharge Symptom Experience Risk Factor Questionnaire for COVID-19 Patients | up to 20 weeks
  The investigators used the Post Discharge Experience Assessment Questionnaire for COVID-19 Patients and the Post Discharge Symptom Experience Risk Factor Questionnaire for COVID-19 Patients were used.Stratified random sampling was used to conduct a cross-sectional survey of 384 patients in recovery from COVID-19.Exploratory factor analysis was used to determine the cluster of symptoms, and a binary logistic regression analysis was used to identify the risk factors associated with this symptom cluster.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No